CLINICAL TRIAL: NCT05636228
Title: Phase 2, Multicenter, Randomized, Double-Masked, Vehicle-Controlled Study of INV-102 Ophthalmic Solution in Patients With Acute Infectious Keratoconjunctivitis
Brief Title: Study of INV-102 Ophthalmic Solution in Adults With Acute Infectious Keratoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Invirsa, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INV-102-CS-002
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Acute Infectious Keratoconjunctivitis
Keywords: pink eye; conjunctivitis
MeSH Terms: conditions — Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INV-102 0.7% Three Times per Day (TID) (Experimental): INV-102 ophthalmic solution administered for about 1 week
  Interventions: Drug: INV-102
- Vehicle TID (Placebo Comparator): INV-102 ophthalmic solution administered for about 1 week
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: INV-102 — INV-102 Ophthalmic Solution
  Arms: INV-102 0.7% Three Times per Day (TID)
Drug: Vehicle — Vehicle Ophthalmic Solution
  Arms: Vehicle TID

SUMMARY:
Phase 2, randomized study to assess topically administered eyedrops of INV-102 compared to vehicle during 1-week dosing in participants with Acute Infectious Keratoconjunctivitis (AIK). Participants will return for a follow up visit 1 week after end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥ 18 years of age
* A clinical diagnosis of AIK with a minimum of a 2+ (moderate) conjunctival hyperemia and a minimum of 1+ (mild) discharge (whether it be watery or purulent) in at least one eye

Exclusion Criteria:

* Untreated keratoconjunctivitis of any type that has lasted 96 consecutive hours or more prior to baseline visit
* Infectious blepharitis as the primary cause of ocular hyperemia and discharge in the opinion of the investigator (Note: If the blepharitis is secondary to the conjunctivitis, the patient can be included)
* Suspected allergic conjunctivitis as a primary cause of conjunctival hyperemia (bulbar redness) and/or discharge in the opinion of the Investigator
* Suspected corneal ulcer
* Ocular topical steroid use within two weeks prior to baseline visit
* Ocular topical antibiotic use for less than 24 hours or greater than 96 hours of dosing prior to Baseline visit (this does NOT exclude naïve patients or patients that have not taken topical antibiotics)
* Ocular topical povidone iodine use within 1 week prior to baseline visit
* Systemic antibiotic use within 2 weeks prior to baseline visit
* Ocular topical or systemic anti-fungal within 2 weeks prior to baseline visit
* Ocular topical or systemic anti-viral use within 2 weeks prior to baseline visit
* Corticosteroid (including but not limited to oral, intranasal, inhaled, topical, etc.) or any immunosuppressant use within 30 days prior to Baseline visit
* On current treatment for herpes keratitis (evidence of herpes keratitis and/or ocular dendrites can be included)
* Known or suspected ocular fungal infection or ocular microsporidia infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
To Evaluate the Change in Combined Clinical Score | Through End of Treatment (Day 8)
  To evaluate the efficacy of INV-102 compared to vehicle control in reducing Combined Clinical Score (bulbar hyperemia plus conjunctival discharge) in patients with AIK. Conjunctival hyperemia will be rated by using the modified version of Cornea and Contact Lens Research Unit grading scale for bulbar redness, which ranges from 0 (none) to 4 points (very severe). Conjunctival discharge will be assessed using the chart below from Schwab and Friedlander (2002) to score conjunctival discharge from 0 (absent/normal) to 3 (severe).

SECONDARY OUTCOMES:
To Evaluate the Percent of participants requiring rescue | Day 3
  To evaluate the percent of patients requiring rescue therapy from Day 3 in the INV-102 arm compared to vehicle control

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - Global Research Management, Glendale, California
  - Foothill Eye Institute, Pasadena, California
  - Shettle Eye Research, Largo, Florida
  - D & H National Research Centers, INC, Miami, Florida
  - My Community Research Center, Inc., Miami, Florida
  - Quantum Clinical Trials, Miami Beach, Florida
  - Kannarr Eye Center, Pittsburg, Kansas
  - Oculos Clinical Research, Garner, North Carolina
  - Athens Eye Care, Athens, Ohio
  - Revolution Research/ Lake Travis Eye and Laser Center, Lakeway, Texas
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Mahidol university, Bangkok